CLINICAL TRIAL: NCT01426594
Title: Real-life Experience of the Use of Isomers as METPURE XL (S (-) Metoprolol Succinate) for Evaluation of Efficacy, Safety and Tolerability in the Management of Cardiovascular Disease in Colombian Patients
Acronym: XPERT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Closter Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: COL-CARDIO-NIS002
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension; Coronary Disease
Keywords: Observational; Colombia; Metpure XL
MeSH Terms: conditions — Hypertension; Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a Phase 4, observational, open study in patients who their doctor has prescribe METPURE XL (S (-)metoprolol succinate)by clinical practice. No medication was provided by the sponsor. The planned observation time is 8 weeks. The 8 weeks of observation involves an evaluation of baseline followed by information gathered from the assessment visits at week 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were prescibed with s(-)metoprolol succinate(25mg, 50mg), depending on their clinical condition and use locally approved will be eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care adults
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Effect of therapy in the management of cardiovascular diseases | 8 weeks
  The objective is to mesure the effect of Metpure XL in cadiovascular diseases as hypertension, post MI and coronary disease

SECONDARY OUTCOMES:
Evaluate and compare the rate of compliance with treatment | 8 weeks
  Evaluate the compliance with METPURE XL, to be able to identify possible reasons for noncompliance or quitting the treatment
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
  To assess the safety pattern in Colombian subjects using s(-)metoprolol succinate

CONTACTS AND LOCATIONS:
Locations (1):
- Country Club de Bogota, Bogotá, Colombia